CLINICAL TRIAL: NCT07046039
Title: The Impact of Untreated Depression and Anxiety in Patients With Skin Diseases: A Cross-sectional Study in Jeddah
Brief Title: The Impact of Untreated Depression and Anxiety Among Patients With Skin Diseases in Jeddah, Saudi Arabia.
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Hadeel Omar Aljohani, Medical student Researcher, King Abdulaziz University
Other Study IDs: 703-23
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Alopecia Areata; Acne Vulgaris; Psoriasis; Atopic Dermatitis (Eczema); Rosacea; Hidradenitis Suppurativa (HS); Vitiligo
Keywords: Psychodermatology; Untreated mental health
MeSH Terms: conditions — Alopecia Areata; Acne Vulgaris; Psoriasis; Dermatitis, Atopic; Eczema; Rosacea; Hidradenitis Suppurativa; Vitiligo

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the prevalence and severity of untreated depression and anxiety among adults with skin diseases in Jeddah, Saudi Arabia. The main question it aims to answer is:

Do patients with skin diseases experience significant levels of untreated depression and anxiety?

Participants diagnosed with skin conditions such as acne, eczema, or psoriasis completed the PHQ-9 and GAD-7 questionnaires to assess their mental health symptoms. The study also explores whether factors like age or type of skin disease are associated with more severe psychological distress.

DETAILED DESCRIPTION:
This cross-sectional observational study was conducted to assess the prevalence and severity of untreated depression and anxiety among adult patients diagnosed with common dermatological conditions in Jeddah, Saudi Arabia. The study focused on patients living with acne vulgaris, atopic dermatitis (eczema), psoriasis, vitiligo, rosacea, hidradenitis suppurativa, and alopecia. Conditions that are not only physically distressing but also associated with significant psychological impact.

Participants were recruited through dermatology clinics and online platforms. Standardized and validated screening tools, including the Patient Health Questionnaire-9 (PHQ-9) and the Generalized Anxiety Disorder-7 (GAD-7), were used to evaluate symptoms of depression and anxiety. Participants were eligible if they were between 18-65 years old, residing in Jeddah, and had not received prior psychiatric treatment for depression or anxiety.

The study also examined potential correlations between psychological distress and clinical or demographic variables such as age, sex, income level, education, and disease severity. Statistical analyses were conducted to identify significant predictors of untreated mental health symptoms in this population.

By quantifying the emotional burden associated with skin disease and identifying at-risk subgroups, the study aims to support the integration of routine mental health screening into dermatologic practice. The findings underscore the need for a more comprehensive, biopsychosocial approach to dermatology care in Saudi Arabia, where psychological symptoms are often underrecognized and undertreated.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adults aged 18 to 65 years
  2. Residents of Jeddah, Saudi Arabia
  3. Diagnosed with one or more of the following skin diseases: acne vulgaris, atopic dermatitis (eczema), psoriasis, vitiligo, rosacea, hidradenitis suppurativa, or alopecia areata
  4. Able to complete the study questionnaire in Arabic or English
* Exclusion Criteria:

  1. Age below 18 or above 65 years
  2. Absence of diagnosis for the specified skin diseases
  3. Presence of chronic systemic illnesses such as diabetes, cardiovascular diseases, hypertension, or epilepsy
  4. Inability to provide informed consent or complete the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years residing in Jeddah, Saudi Arabia, who have been diagnosed with one or more of the following dermatological conditions: acne vulgaris, atopic dermatitis (eczema), psoriasis, vitiligo, rosacea, hidradenitis suppurativa, or alopecia areata. Participants were recruited from dermatology outpatient clinics and through online social media platforms.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of untreated anxiety | 1 day (Assessed at one point in time during the study.)
  The proportion of patients with dermatological conditions who score above the clinical threshold for anxiety on the Generalized Anxiety Disorder-7 (GAD-7) scale.
Prevalence of untreated depression | 1 day (Assessed at one point in time during the study.)
  The proportion of patients with dermatological conditions who score above the clinical threshold for depression on the Patient Health Questionnaire-9 (PHQ-9).

SECONDARY OUTCOMES:
Correlation between skin disease severity and psychological distress | 1 day (Assessed at one point in time during the study.)
  Statistical assessment of the relationship between the severity of skin diseases (categorized as mild, moderate, or severe) and the levels of depression and anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University - Faculty of Medicine, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Although aggregate study results will be published, individual participant data (IPD) will not be shared because no identifiable data was collected, ensuring participant privacy and confidentiality.